CLINICAL TRIAL: NCT01637597
Title: An Exploratory Study Of Crizotinib Efficacy In Non-Small Cell Lung Cancer Patients With Anaplastic Lymphoma Kinase Translocation Determined By Different Molecular Diagnostic Methods
Brief Title: Crizotinib Efficacy In Non-Small Cell Lung Cancer Patients With Anaplastic Lymphoma Kinase Translocation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201204080RIC
Record Dates: First submitted 2012-06-28; First posted 2012-07-11 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Non-small Cell Lung Cancer(NSCLC)
Keywords: Non-small cell lung cancer(NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tumor tissue are being collected during the course of this study, to assess the safety and tolerability and spectrum of side effects of the study drug. However, it is possible that after completion of all study-related analyses, some volume of samples may remain. These left-over samples could be a valuable resource for future research.
  Before any left-over samples can be used for any research other than that specified in the protocol, patient must sign an additional future use consent from indicating they give their permission for these samples to be used in future research. By signing the main consent form, patients are only giving their permission to use their samples for the study related procedures.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an exploratory study in patients with locally advanced or metastatic Non-small cell lung cancer. Patients who are eligible to apply for Extended Access Program of crizotinib must have ALK translocation detected by RT-PCR, IHC or FISH analyses methods.

DETAILED DESCRIPTION:
This is an exploratory non-randomized study in patients with locally advanced or metastatic NSCLC. Patients who are eligible to apply for Extended Access Program of crizotinib must have ALK translocation detected by RT-PCR, IHC or FISH analyses methods. Patients who failed and progressed through at least one line of platinum containing chemotherapy and who are older than 70 years old with failure of chemotherapy will be eligible for this study. We will screen EML4-ALK fusion gene by RT-PCR (HotSart Taq Master Mix Kits, Qiaqen) from patients' malignant pleural effusions and the detail was described in previous study[1]. We will also use IHC analyses (5A4 monoclonal antibody, Novocastra) to screen ALK protein expression in patients' FFPE tumor sections. We will further do FISH analysis by using commercial Vysis LSI ALK Dual Color, Break Apart Rearrangement Probe (2p23) (Abott Molecular Inc., Des Plaines, IL) to detect ALK rearrangement in positive screening tumors. Samples are deemed to be FISH-positive if more than 15% of 50 scored tumor cells had split ALK 5' and 3' probe signals or had isolated 3' signals[5]. Patients who have ALK rearrangement determined in any of 3 molecular analyses methods and apply for crizotinib will receive 250mg of crizotinib twice daily until disease progression, unacceptable toxicities or the withdrawal of consent is noted.

Patients will be monitored carefully for the development of adverse experiences. Adverse experiences will be evaluated according to criteria outlined in the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Patients will also be monitored for clinical and/or radiographic evidence of disease progression according to RECIST 1.1.

The primary endpoint of the study is overall response rate in patients with positive ALK determined from different molecular analysis methods. The secondary endpoint included overall response in specific subsets of patients, progression-free survival (PFS), and overall survival (OS) at 1 year. PFS is defined as the time from day 1 of crizotinib to disease progression or patient's death. OS was defined as the time from day 1 of crizotinib treatment to patient's death.

During the treatment, patients will have safety measurements performed at specified time points. Disease response will be assessed during the study by radiographic (e.g., CT or MRI), and clinical (e.g., physical examination) evaluations, if applicable. Overall tumor response will be assessed at the designated time points (every 12 weeks, using Response Evaluation Criteria in Solid Tumors (RECIST, Version 1.1). The crizotinib treatment could be continued after RECIST-defined disease progression if clinical benefit is still noted by primary physician.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have locally advanced or metastatic NSCLC (Stage IIIb or Stage IV by AJCC 7th.) with positive ALK determined by RT-PCR or IHC (5A4, 3+ score). Patients must have failed and progressed through at least one line of platinum containing chemotherapy or failed and progressed through chemotherapy if they were older than 70 years old.
2. Patient must have at least one measurable lesion.
3. Patient is male or female and ≥ 20 years of age on the day of signing informed consent.
4. Patient must have performance status ≤ 2 on the ECOG Performance Scale.
5. Patient must have adequate organ function as indicated by the following laboratory values: adequate liver (total bilirubin < 1.5 x the upper limit of normal (ULN), total bilirubin > 1.5 x ULN but biliary obstruction is documented radiologically, transaminases < 2.5 x ULN or < 5 x ULN if due to liver metastases), renal (creatinine < 2 x ULN) and bone marrow function (hemoglobin > 8g/dL, absolute neutrophil count > 1 X 109/L and platelets > 30 X 109/L)
6. Female patient of childbearing potential has a negative serum or urine pregnancy test β-hCG within 5 days prior to receiving the first dose of study medication.
7. Patients have completed chemotherapy regimens have residual toxicity < Grade 1 except alopecia.
8. Patient, or the patient's legal representative, has voluntarily agreed to participate by giving written informed consent.
9. Patient is able to swallow capsules and has no surgical or anatomical condition that will preclude the patient from swallowing and absorbing oral medications on an ongoing basis.

Exclusion Criteria:

1. Patient who has had chemotherapy within 2 weeks prior to Day 1 of Cycle 1 or has not recovered from the adverse events due to previous agents prior to Day 1 of Cycle 1. If the patient has residual toxicity from prior treatment, toxicity must be ≤ Grade 1 except alopecia.
2. Patient who has had major surgery within 4 weeks prior to starting of treatment or expect major surgery in the study duration. Patient who has had prior radiotherapy (except brain) within 1 week prior to Day 1 of Cycle 1.
3. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days, or 5x half-life from prior agents, whichever is longer, of Day 1 of this study.
4. Patient has known active CNS metastases and/or carcinomatous meningitis unless patients were clinically stable for 2 weeks after radiotherapy.
5. Patient with a primary central nervous system tumor.
6. Patient has known hypersensitivity to the components of study drug or its analogs.
7. Patient has severe systemic disease.
8. Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
9. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
10. Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse.
11. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
12. Patient is known to be Human Immunodeficiency Virus (HIV)-positive
13. Patient currently has active Hepatitis B which is defined as patient has positive serum HBsAg with ALT > 2 x ULN and HBV DNA > 20,000 IU/mL.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic NSCLC who are eligible to apply for Extended Access Program of crizotinib must have ALK translocation detected by RT-PCR, IHC or FISH analyses methods.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate in patients with positive ALK determined from different molecular analysis methods. | It is defined as the time from day 1 of crizotinib to disease progression or patient's death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
Overall survival (OS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James Chih-Hsin Yang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin YT, Yu CJ, Yang JC, Shih JY. Anaplastic Lymphoma Kinase (ALK) Kinase Domain Mutation Following ALK Inhibitor(s) Failure in Advanced ALK Positive Non-Small-Cell Lung Cancer: Analysis and Literature Review. Clin Lung Cancer. 2016 Sep;17(5):e77-e94. doi: 10.1016/j.cllc.2016.03.005. Epub 2016 Mar 30. PMID 27130468
- [Derived] Lin YT, Wang YF, Yang JC, Yu CJ, Wu SG, Shih JY, Yang PC. Development of renal cysts after crizotinib treatment in advanced ALK-positive non-small-cell lung cancer. J Thorac Oncol. 2014 Nov;9(11):1720-5. doi: 10.1097/JTO.0000000000000326. PMID 25436806